CLINICAL TRIAL: NCT00485225
Title: An Open-Label, Two-Stage, Phase II Study to Explore the Titration Schedule for Transitioning Opioid-Experienced Patients With Non-Malignant Moderate to Severe Chronic Pain From Current Opioid Therapy to EN3270.
Brief Title: Open Label, Safety Study of EN3270 in Patients With Moderate to Severe Non-malignant, Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3270-201
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2011-12

CONDITIONS: Chronic, Non Malignant Pain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Transdermal patch (EN3270) - Titration 1 (Experimental)
  Interventions: Drug: EN3270
- Transdermal patch (EN3270) - Titration 2 (Experimental)
  Interventions: Drug: EN3270
- Transdermal patch (EN3270) - Titration 3 (Experimental)
  Interventions: Drug: EN3270
- Transdermal patch (EN3270) - Titration 4 (Experimental)
  Interventions: Drug: EN3270

INTERVENTIONS:
Drug: EN3270 — Transdermal Therapeutic System

SUMMARY:
Two stage study looking at different titration schedules in patients with moderate to severe non-malignant chronic pain. Up to 80 patients at approximately 15 centers in the US to be enrolled. Study participation is approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Opioid experienced
* Hx (min 3 months) of moderate to severe pain of non-malignant that is well controlled with current pain therapy
* On a stable dose of opioid medication for greater than or equal to 14 days
* Have an adequate personal support system including a co-habitant
* Are able and willing to follow verbal and written instructions and provide written informed consent

Exclusion Criteria:

* Are pregnant or lactating
* Have pain secondary to a confirmed or suspected neoplasm
* Have a history or physical examination finding incompatible with safe participation in the study
* Have a history of alcohol or drug abuse
* Have a history or physical examination finding of clinically significant skin abnormalities that would preclude use of a transdermal patch (e.g., psoriasis)
* Have a history of or currently manifesting a clinically significant psychiatric disorder
* Have a known history of allergy that negatively impacts respiratory function to a clinically significant level
* Plan to have an MRI while on the study
* Have any clinically significant condition that would, in the opinion of the investigator, preclude safe study participation
* Are scheduled for surgery requiring general anesthesia within the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety and minimum titration period | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Clinical Research, Berlin, New Jersey, United States